CLINICAL TRIAL: NCT06575309
Title: Longitudinal Study of the in Vitro Action of Low Molecular Weight Heparin (LMWH) in Pregnant Women by Thrombinography
Brief Title: THROmbinography in Pregnant Woman and in Vitro Action of Low Molecular Weight HEparin
Acronym: TROPHE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RBHP 2024 LEBRETON; 2024-A00109-39 (Other: ANSM)
Record Dates: First submitted 2024-07-22; First posted 2024-08-28 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-05

CONDITIONS: Pregnant Women; Venous Thromboembolic Disease
Keywords: Thrombography; Pregnancy; Postpartum; Low molecular weight heparins (LMWH)
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women
  Interventions: Biological: Blood test

INTERVENTIONS:
Biological: Blood test — The procedures added as part of this research are 6 blood samples, the volumes of which do not exceed the volume authorized in the order of February 17, 2021, i.e. 27mL.

SUMMARY:
Pregnancy is associated with major changes affecting all satges of hemostasis. Certain procoagulant factors are increased, such as factors VII, VIII, IX, X, XII, fibrinogen and Von Willebrand factor. Anticoagulant molecules are also affected by pregnancy, notably the protein C - protein S (PC - PS) system. overall, PC activity is little affected by pregnancy, increasing in the 2nd trimester and decreasing in the 3rd, but remaining within normal values. PS decreases from the first trimester of pregnancy, then progressively with gestational age. Antithrombin is stable during pregnancy.

The increased in most coagulation factors, combined with the decrease in concentrations of anticoagulant molecules, creates a state of relative hypercoagulability that protects women from bleeding during homostatic challenge of childbirth, but predisposes them to venous thromboembolic events.

The risk of venous thromboembolism (VTE) during pregnancy is increased compared to non-pregnant women of the same age. The post-partum period is also considered a thrombotic risk state for up to 12 weeks after delivery. Data on the incidence of VTE as a function of gestational age are contradictory: depending on the study, incidence may be stable or increase with advancing pregnancy.

Low-molecular-weight heparin (LMWH) is the anticoagulant treatment of choice for prophylactic or curative treatment of VTE during pregnancy.

Physiological changes during pregnancy may alter the pharmacokinetic properties of LMWH. The increased volume of distribution and higher glomerular filtration rate may result in a reduced anticoagulant effect. On the other hand, the state of hypercoagulability probably counteracts the anticoagulant effect of LMWH. Nevertheless, the need to adjust doses during pregnancy remains controversial, and monitoring of anti-Xa activity is not clearly recommended. The optimal dose of LMWH in pregnant women, for both preventive and curative treatment, remains poorly understood. Initiation of treatment with LMWH therefore requires discussion of the dosage to be administered.

Assessment of anticoagulation using more precise tools than those currently available on a routine basis could be useful in this context.

Thrombinography enables the amount of thrombin generated in the presence of coagulation activators to be assessed over time. This tool can be used to assess the impact of in vitro addition of different doses of LMWH in pregnant versus non-pregnant women and in the postpartum period.

In this pilot study, the investigators propose to evaluate thrombin generation, before and after in vitro addition of LMWH, in pregnant women longitudinally, during the 3 trimesters of pregnancy, postpartum and post-pregnancy.

DETAILED DESCRIPTION:
Pregnancy is considered a risk factor for venous thromboembolism (VTE), with deep vein thrombosis and pulmonary embolism the main causes of maternal morbidity and mortality. studies report a 5-fold increase in risk during pregnancy. The post-partum period is also at risk of thrombosis, with 24.4 events per 100,000 births observed in the first 6 weeks after delivery, compared with 2.3 in the same period a year later. During the period 7 to 12 weeks after delivery, the risk is modest but still significant. Pregnant women are therefore at high risk of thrombosis during the first 6 weeks post-partum. This risk decreases, but persists for up to 3 months. Although many data suggest that the incidence of VTE is similar during the 3 trimesters of pregnancy, a recent study actually shows that the risk increases exponentially throughout gestation.

Treatment with low-molecular-weight heparin (LMWH) is the anticoagulant treatment of choice for the prevention or cure of VTE during pregnancy, and throughout the 3 trimesters of gestation, due to its ease of administration and monitoring, and the low incidence of adverse effects.

However, physiological changes during pregnancy may alter the pharmacokinetic properties of LMWH. The increased volume of distribution and higher glomerular filtration rate may result in a reduced anticoagulant effect. Nevertheless, the need to adjust doses during pregnancy remains controversial. Some authors suggest simply increasing the dose according to weight, especially at therapeutic doses. Others go further, advocating dose adjustment not only according to weight, but also by monitoring anti-Xa activity to keep it within defined limits. On the other hand, other authors have shown that few women require dosage adjustment.

As a result, monitoring of anti-Xa activity is not clearly recommended, and the true hemostatic profile of women undergoing LMWH treatment is still open to question. This means that the optimal dose of LMWH in pregnant women, for both preventive and curative treatment, remains poorly understood. Initiation of treatment with LMWH therefore requires discussion of the dosage to be administered, in order to avoid over- or under-dosing and the inherent risks. For prophylaxis, a single daily dose of LMWH (e.g. enoxaparin 40 mg) is commonly administered throughout pregnancy, without monitoring anti-Xa activity and without taking into account physiological changes during pregnancy.Recently, Bistervels et al. recommended the use of low-dose LMWH for the prevention of deep vein thrombosis. Nevertheless, it appears that intermediate doses adapted to weight may be justified in women with a body mass index of less than 30, to prevent pulmonary embolism or in the post-partum period . Anticoagulation assessment using more precise tools than those currently available on a routine basis could be useful in this context.

There is a lack of data on the true state of hypercoagulability and the mechanisms involved during pregnancy. Most studies have focused on the levels of procoagulant and anticoagulant factors. This type of study gives only a fragmentary view of the haemostatic balance of pregnant women. More recently, more comprehensive coagulation tests such as thrombinography have been used in pregnant women.

The purpose of plasma coagulation is to generate a large quantity of thrombin, the key coagulation enzyme, enabling fibrinogen to be converted into a fibrin network. Routine coagulation tests (PT, APTT) use supra-physiological doses of coagulation activators, and report only the first traces of fibrin in plasma, corresponding to less than 5% of the thrombin formed in vivo. Conventional tests therefore fail to study the kinetics of the remaining 95% of thrombinoformation. The C.A.T. (Calibrated Automated Thrombography) method was developed by Hemker and is distributed by Stago®.

Thrombinography thus enables us to monitor thrombin generation kinetics, integrating the action of procoagulant and anticoagulant factors, unlike standard haemostasis tests (PT and APTT). As a result, measuring thrombin generation better reflects a subject's hemostatic potential, especially when the subject presents complex variations in coagulation molecules, as is the case during pregnancy. Available data on thrombinography in pregnancy are limited and contradictory. Some authors consider that thrombin generation increases as early as the first trimester of pregnancy and then remains stable throughout pregnancy, whereas others find an increase during pregnancy, at least during the first 2 trimesters. There are few longitudinal studies evaluating thrombin generation during pregnancy and post-partum in a given pregnant woman. These studies are carried out on small numbers.

A global coagulation test such as thrombinography could be used to assess the impact of in vitro addition of different doses of LMWH in pregnant and postpartum women.

Preliminary dose-ranging studies carried out in the laboratory have shown that the in vitro addition of LMWH corresponding to 0.3 IU/mL anti-Xa activity results in a decrease in thrombinography parameters. The area under the curve, or AUC, was reduced by 50%. Comparing thrombin generation profiles with and without in vitro addition of LMWH in pregnant versus non-pregnant women can help assess the action of LMWH. Indeed, some authors have studied the effect on thrombin generation of in vitro addition of LMWH to the plasma of pregnant and non-pregnant women. In vitro addition of LMWH reduces thrombin generation in pregnant and non-pregnant women, but the percentage of inhibition is significantly lower in pregnant women, reflecting a "resistance" to the action of LMWH. Nevertheless, the population studied was small (n=12), and anti-Xa activity was not determined. What's more, only women in their first trimester of pregnancy were included, so this study does not allow longitudinal assessment of resistance during pregnancy and post-partum.

In this pilot study, the investigators propose to evaluate thrombin generation, before and after in vitro addition of LMWH, in pregnant women longitudinally, during the 3 trimesters of pregnancy, post-partum and post-pregnancy.

This descriptive study could be the indispensable preamble to a larger-scale clinical study aimed at using thrombinography to optimize anticoagulant therapy in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Normal 1st trimester pregnancy
* Age > 18

Exclusion Criteria:

* Coagulation disease (Von Willebrand disease, known coagulation factor deficiency before pregnancy)
* VTE history
* First-degree family history of idiopathic VTE
* Known biological risk factor for thrombosis Inherited deficiencies in coagulation inhibitors (antithrombin, protein C, protein S) Factor V Leiden polymorphism Prothrombin gene 20210G>A polymorphism Anti-phospholipid antibodies
* Current anticoagulant use (VKA, heparins, etc.)
* Gestational diabetes detected in the 1st trimester
* Pre-existing type 1 and type 2 diabetes
* History of pathological pregnancy Premature delivery Postpartum hemorrhage Preeclampsia
* Hepatopathy
* Obesity (BMI ≥ 30)
* Infections (HIV, HBV, HCV...)
* Autoimmune diseases
* Pregnancy resulting from in vitro fertilization protocol
* Multiple pregnancy
* Patient under guardianship, curatorship or safeguard of justice
* Patient not covered by a social security scheme
* Patient deprived of liberty

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with no health problems recruited during their 1st trimester of pregnancy, then monitored throughout the pregnancy.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
The endogenous thrombin potential | through study completion, an average of 1 year
  Thrombinography provides a graphical representation of the amount of thrombin generated as a function of time (thrombinogram). The "endogenous thrombin potential (ETP)" corresponds to the area under the curve, reflecting the overall quantity of thrombin generated (in nM.min-1).LMWH inhibition of PTE is expressed as the inhibition ratio: (basal PTE - PTE with LMWH)/basal PTE.

SECONDARY OUTCOMES:
The lag time | through study completion, an average of 1 year
  This is the latency time before the start of thrombin generation (in min).Inhibition of lag time by LMWH is expressed as the inhibition ratio: (basal lag time - lag time with LMWH)/basal lag time.
the peak Height | through study completion, an average of 1 year
  This is the maximum thrombin concentration (in nM thrombin) (Cmax). Inhibition of this concentration by LMWH is expressed as the inhibition ratio: (basal peak heigh - peak heigh with LMWH)/basal peak heigh.
The time to peak | through study completion, an average of 1 year
  This is the time after which the maximum amount of thrombin is reached (in min). Inhibition of time to peak by LMWH is expressed as an inhibition ratio: (basal Time to peak - Time to peak with LMWH)/basal Time to peak.
The start tail | through study completion, an average of 1 year
  This is time after which no more thrombin is generated (in min). Inhibition of start tail by LMWH is expressed as an inhibition ratio: (basal start tail - start tail with LMWH)/basal start tail.
The "velocity index" | through study completion, an average of 1 year
  This is the thrombin generation rate (in nM.min). Inhibition of velocity index by LMWH is expressed as an inhibition ratio: (basal velocity index - velocity index with LMWH)/basal veocity index

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien Lebreton, Principal Investigator — CHU de Clermont-Ferrand
Locations (2):
- France (2):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU Estaing, Clermont-Ferrand